CLINICAL TRIAL: NCT00364546
Title: A Randomized, Double-Blind, Active-Control, Parallel-Group, 90-Day Safety Study of CG5503 Immediate Release (IR) or Oxycodone IR in Subjects With Chronic Pain From Low Back Pain or Osteoarthritis of the Hip or Knee
Brief Title: A Study to Evaluate 90-Day Safety of Tapentadol(CG5503) Immediate Release (IR) or Oxycodone Immediate Release in Patients With Chronic Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: Grünenthal GmbH (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR011212
Record Dates: First submitted 2006-08-11; First posted 2006-08-15 (Estimated); Last update posted 2011-06-09 (Estimated); Status verified 2010-04

CONDITIONS: Osteoarthritis; Pain Intensity Assessment; Arthralgia; Sciatica; Low Back Pain
Keywords: Osteoarthritis; Pain; Low Back Pain; Hip Pain; Knee Pain; Backache; tapentadol
MeSH Terms: conditions — Osteoarthritis; Arthralgia; Sciatica; Low Back Pain; Pain; Back Pain

INTERVENTIONS:
Drug: CG 5503;tapentadol

SUMMARY:
The purpose of this study is to evaluate the safety of CG5503 base Immediate Release(IR) 50 mg or 100 mg taken every 4 to 6 hours as needed over the long-term exposure of 90 days in patients who have chronic pain.

DETAILED DESCRIPTION:
CG5503 is a centrally active pain-relieving drug being investigated for the treatment of acute and chronic pain. This study is designed to assess the safety of CG5503 Immediate Release (IR) in men and women who are 18 years of age or older and who have had chronic (for at least 3 months) low-back pain or chronic pain from osteoarthritis of the hip or knee, and who require daily analgesic medication. In this double blind study (neither patients nor investigators will know what treatment is given), patients will be randomly (patients are assigned different treatments based on chance) assigned to receive either CG5503 base IR or oxycodone IR to begin a 90 day treatment during which each patient will return to the medical facility every 2 weeks. For the CG5503 IR group, patients will take 50 or 100 mg orally every 4 to 6 hours as needed to a maximum dose of 600 mg per day. Oxycodone IR patients will take 10 or 15 mg orally every 4 to 6 hours as needed to a maximum dose of 90 mg per day. Patients may continue taking their regular, stable, non-opioid medication throughout the study. The effectiveness of study treatment (CG5503 base IR or oxycodone) will be assessed with 11-Point Numerical Rating Scale and Patient Global Impression of Change. Using these scales, patients will indicate their pain intensity level and overall status of their well-being. Opioid withdrawal symptoms of CG5503 IR dose of 50 or 100 mg will be assessed with clinical opioid withdrawal scale [Subjective Opiate Withdrawal Scale (SOWS) and Clinical Opiate Withdrawal Scale (COWS)] at the end of treatment. Using these scales, patients will indicate the physical components of drug withdrawal and the severity of symptoms associated with rapid withdrawal. Safety will be assessed using physical examination, monitoring of adverse events, clinical and laboratory measures, and 12 lead electrocardiogram (ECG) results. Constipation, vomiting, and sleep assessments will be performed. No formal hypothesis testing will be done in this study. For the CG5503 IR group, patients will take a flexible dose of 50 or 100 mg orally every 4 to 6 hours as needed to a maximum dose of 600 mg per day for 90 days. Oxycodone IR patients will take a flexible dose of 10 or 15 mg orally every 4 to 6 hours as needed to a maximum dose of 90 mg per day for 90 days.

ELIGIBILITY:
Inclusion Criteria:

* A clinical diagnosis of one of the following: low-back pain of non-malignant origin for at least 3 months, osteoarthritis of the knee or hip for at least 3 months
* require daily doses of analgesia medication for chronic pain that is consistent with or makes them candidates for treatment at Step 2 or higher of the WHO Pain Relief Ladder
* post-washout baseline pain intensity score >4 on an 11-point numerical rating scale

Exclusion Criteria:

* History of seizure disorder or epilepsy
* uncontrolled hypertension
* currently treated with monoamine oxidase inhibitors
* systemic steroid therapy, excluding inhalers or topical steroids, within 3 months before screening
* history of malignancy within the past 2 years, with the exception of basal cell carcinoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 877 (Actual)
Dates: Start 2006-07; Primary Completion 2007-06 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
The primary outcomes include incidence of adverse events, changes in laboratory measures, results of physical exams, and results of 12-Lead ECG.

SECONDARY OUTCOMES:
The secondary outcomes, among others, include COWS and SOWS assessments; patient assessment of constipation symptoms; vomiting and sleep assessments; pain intensity assessment; patient global impression of change.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Derived] Vorsanger G, Xiang J, Biondi D, Upmalis D, Delfgaauw J, Allard R, Moskovitz B. Post hoc analyses of data from a 90-day clinical trial evaluating the tolerability and efficacy of tapentadol immediate release and oxycodone immediate release for the relief of moderate to severe pain in elderly and nonelderly patients. Pain Res Manag. 2011 Jul-Aug;16(4):245-51. doi: 10.1155/2011/323985. PMID 22059194
- [Derived] Hale M, Upmalis D, Okamoto A, Lange C, Rauschkolb C. Tolerability of tapentadol immediate release in patients with lower back pain or osteoarthritis of the hip or knee over 90 days: a randomized, double-blind study. Curr Med Res Opin. 2009 May;25(5):1095-104. doi: 10.1185/03007990902816970. PMID 19301989
- See also: A Randomized, Double-Blind, Active-Control, Parallel-Group, 90-Day Safety Study of CG5503 (Tapentadol HCl) Immediate Release or Oxycodone Immediate Release in Subjects With Chronic Pain From Low Back Pain or Osteoarthritis of the Hip or Knee — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=726&filename=CR011212_CSR.pdf